CLINICAL TRIAL: NCT03572985
Title: Development of Assessment Method for Driving Ability Using Driving Simulator in Healthy Volunteers #3: Alcohol Calibration
Brief Title: Development of Assessment Method for Driving Ability Using Driving Simulator in Healthy Volunteers #3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nagoya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: DS-204-03; JapicCTI-184006 (Other: JapicCTI)
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2019-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Blood alcohol concentration (BAC) level 0.025 % (Other): Drink beverages containing alcohol calculated to have a blood alcohol concentration of 0.025%
  Interventions: Other: Road-tracking test; Other: Car-following test; Other: Harsh-braking test
- BAC level 0.05 % (Other): Drink beverages containing alcohol calculated to have a blood alcohol concentration of 0.05%
  Interventions: Other: Road-tracking test; Other: Car-following test; Other: Harsh-braking test
- BAC level 0.09 % (Other): Drink beverages containing alcohol calculated to have a blood alcohol concentration of 0.09%
  Interventions: Other: Road-tracking test; Other: Car-following test; Other: Harsh-braking test
- BAC level 0 % (Other): Drink beverages containing non alcohol
  Interventions: Other: Road-tracking test; Other: Car-following test; Other: Harsh-braking test

INTERVENTIONS:
Other: Road-tracking test — Driving with simulator program for SDLP measurement
Other: Car-following test — Driving with simulator program for DCV measurement
Other: Harsh-braking test — Driving with simulator program for BRT measurement

SUMMARY:
The purpose of this study is to collect alcohol calibration data for the driving simulator.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 and <25.0 kg/m^2 at screening inspection
* No visual impairment (enable to correct the vision with eyeglasses or contact lens)
* Receive a prior explanation on the study, able to accept its content, and capable to provide voluntary written consent for participation in this study

Exclusion Criteria:

* History of drug and food allergy
* Alcohol dependence, drug dependence or abnormal drunken (including past history)
* Inappropriate for enrollment in this study was judged by principal investigator or subinvestigator

Ages: 21 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) | 60 min

SECONDARY OUTCOMES:
Distance Coefficient of Variation (DCV) | 5 min
Brake Reaction Time (BRT) | 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Okuyama, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Fukuoka, Japan

REFERENCES:
- [Derived] Iwata M, Iwamoto K, Omura T, Ando M, Ozaki N. Protocol for the development and validation of a driving simulator for evaluating the influence of drugs on driving performance. Medicine (Baltimore). 2019 Feb;98(8):e14613. doi: 10.1097/MD.0000000000014613. PMID 30813188